CLINICAL TRIAL: NCT06926270
Title: Effectiveness of Transcranial Magnetic Stimulation Treatment in Patients Diagnosed With Postpolio Syndrome: A Randomized Controlled Double-Blind Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Arzu On, Prof.Dr, Ege University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1174637
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Postpolio Syndrome
Keywords: Postpolio; poliomyelit; TMS; rTMS; gait speed
MeSH Terms: conditions — Postpoliomyelitis Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SHAM (Sham Comparator): 5 sessions per week; 2 weeks, 90% RMT (resting motor threshold), 1 Hz, 15 min TMS will be applied, but treatment During the procedure, the application head of the device is turned in the opposite direction so that the patient receives TMS treatment.
  effect, but you hear the operating sound of the device and will spend it in the laboratory
  Also, home exercise program:
  quadriceps strengthening and knee isometric exercises
  Interventions: Device: TMS
- INTERVENTION (Experimental): 5 sessions/week, 2 weeks, 90% RMT (resting motor threshold), 1 Hz, 15 min TMS application to patients As the application point, the Cz point on the EEG map, contralateral to the affected extremity, will be taken
  Also, home exercise program:
  quadriceps strengthening and knee isometric exercises
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — Magstim ,Rapid 2

SUMMARY:
The study is planned to include a minimum of 26 patients with paralytic poliomyelitis who meet the PPS diagnostic criteria (1). Patients will be randomized into two groups, and one group will receive only the exercise therapy used in standard treatment, while the other group will receive Transcranial Magnetic Stimulation (TMS) therapy in addition to exercise. TMS will be applied to the study group 5 times a week for 2 weeks, for a total of 10 sessions. The protocol to be applied during the study will be set to 1 Hz, and each session will last 15 minutes. All participants will be evaluated with muscle strength (manual muscle testing), 6-minute walking test, polio-related problems inventory, VAS pain, VAS fatigue, fatigue severity scale, Beck Depression Inventory, Nottingham health profile scales before, at the end of treatment, and at the end of the 3rd month. As a result of the evaluation, the potential positive effects of TMS on patients with PPS will be measured and evidence-based data for the use of this treatment modality in patients with PPS will be obtained. This study will be the first to evaluate the effectiveness of TMS in a controlled manner in a patient group with PPS. As a result of the evaluation, the potential positive effects of TMS on patients with PPS will be measured and evidence-based data will be obtained for the use of this treatment modality in patients with PPS.

ELIGIBILITY:
Inclusion Criteria:-Having been diagnosed with PPS (postpolio syndrome) -Having not received TMS treatment before

-

Exclusion Criteria:-History of epilepsy

* Presence of another disease that may be associated with the symptoms
* Inability to ambulate independently
* Presence of a neurological, psychiatric or vision-related problem that may prevent the patient from answering the questionnaires
* Presence of ferromagnetic material implanted in the body
* Organic brain pathology (vascular, traumatic, tumoral, etc.)
* History of use of drugs that lower the seizure threshold (if not receiving antiepileptic treatment)
* Severe or recent heart disease
* Alcoholism
* Pregnancy

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test | 2 weeks
  It is a test used to assess the level of functional exercise or functional capacity. The patient is asked to walk, but not run, in a 25 m long corridor at the highest possible speed without stopping. At the end of 6 minutes, the number of metres walked by the patient is recorded. The 6 min walk test is an evaluation criterion used in routine and clinical research to assess functional capacity in many diseases such as heart failure, general arthrosis, multiple sclerosis.

SECONDARY OUTCOMES:
Self-reported ımpairments in persons with late effects of polio (SIPP) rating scale | 2 weeks
  It consists of 13 items about PRI that the participants might have been bothered during the past 2 weeks: muscle weakness, muscle fatigue, muscle, and/or joint pain during physical activity and at rest, sensory disturbance, breathing difficulties at rest and during physical activity, cold intolerance, general fatigue, sleep disturbances, concentration difficulties, memory difficulties, and mood swings. The respondents are asked to rate each item as; 1: not at all, 2: little, 3: quite a bit 4: extremely, giving a total sum score ranging from 13 to 52 points. A higher score indicates more self-reported impairments
Nottingham health profile (NHP) | 2 weeks
  It consists of 38 items assessing how severe an impact the respondent thinks their health is having on six dimensions: sleep, physical mobility, energy, pain, emotional reactions, and social isolation. Every item has a different weight, depending on the severity of the symptom. The sum of the weighted scores is 100 for each subdimension. Thus, summing all weighted values of every item, the score between 0 and 100 is obtained for each subdimension. The total score was obtained by summing the scores of six subdimensions, giving the values between 0 and 600. Higher scores indicate a greater level of distress
Visual analogue scale (VAS) for pain and fatigue | 2 weeks
  Severity of pain that the participants have had in the past week was evaluated by using visual analogue scale (VAS) on a 10-cm horizontal line where 0-cm represented "no pain" and 10 cm the "worst imaginable pain"
  Severity of fatigue experienced by the participants in the past week was assessed by using VAS on a 10-cm horizontal line where 0-cm represented "not tired at all" and 10-cm "extremely tired"
Manual muscle testing (MMT) | 2 weeks
  Muscle strength of the hip flexors, knee extensors, knee flexors, ankle dorsiflexors, and plantar flexors were measured bilaterally according to the Medical Research Council Scale . A sum score (manual muscle testing [MMT] sum) was obtained by adding the scores of all muscle groups tested (max score: 50)
Fatigue Impact Scale (FIS) | 2 weeks
  Cognitive, functional and fatigue subscales are available and high scores are associated with poor fatigue level
Beck Depression Scale | 2 weeks
  The Beck depression test is used to measure how intensely depressed a person is during a 1-week period.21 questions; each question is scored between 0 and 3. The degree of depression is determined according to the total score (0-9: minimal depression, 10-16: mild depression, 17-29: moderate depression, 30-63: severe depression).

CONTACTS AND LOCATIONS:
Overall Officials: Arzu On, Prof.Dr, Principal Investigator — Ege Universtiy
Locations (1):
- Ege University Faculty of Medicine, Izmir, BORNOVA, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Altas EU, Askin A, Besiroglu L, Tosun A. Is high-frequency repetitive transcranial magnetic stimulation of the left primary motor cortex superior to the stimulation of the left dorsolateral prefrontal cortex in fibromyalgia syndrome? Somatosens Mot Res. 2019 Mar;36(1):56-62. doi: 10.1080/08990220.2019.1587400. Epub 2019 Apr 8. PMID 30955403
- [Background] Klomjai W, Katz R, Lackmy-Vallee A. Basic principles of transcranial magnetic stimulation (TMS) and repetitive TMS (rTMS). Ann Phys Rehabil Med. 2015 Sep;58(4):208-213. doi: 10.1016/j.rehab.2015.05.005. Epub 2015 Aug 28. PMID 26319963
- [Background] Ertekin C, On AY, Kirazli Y, Kurt T, Gurgor N. Motor evoked responses from the thigh muscles to the stimulation of the upper limb nerves in patients with late poliomyelitis. Clin Neurophysiol. 2002 Apr;113(4):478-84. doi: 10.1016/s1388-2457(02)00043-3. PMID 11955992
- [Background] Willen C, Hou L, Stibrant Sunnerhagen K. A very long-term longitudinal follow-up of persons with late effects of polio. Eur J Phys Rehabil Med. 2020 Apr;56(2):155-159. doi: 10.23736/S1973-9087.20.05918-3. Epub 2020 Feb 10. PMID 32043852
- [Background] Latifoglou E, Cinar E, Tanigor G, On AY. Coexistence of fibromyalgia and post-polio syndrome in persons with prior poliomyelitis in Turkey: the relations with symptoms, polio-related impairments, and quality of life. Disabil Rehabil. 2023 Oct;45(21):3511-3518. doi: 10.1080/09638288.2022.2127931. Epub 2022 Sep 28. PMID 36169616